CLINICAL TRIAL: NCT06809842
Title: Analgesic Efficacy of Blocking Nerve to Vastus Lateralis Muscle Versus Lateral Femoral Cutaneous Nerve After Knee Surgeries: A Randomized Trial
Brief Title: Analgesic Efficacy of Blocking Nerve to Vastus Lateralis Muscle Versus Lateral Femoral Cutaneous Nerve After Knee Surgeries
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Sherif Kamal Arafa, Assistant professor of Anesthesiology, Surgical Intensive Care and Pain Management Department, Faculty of Medicine, KafrElsheikh University, KafrElsheikh, Egypt., Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MKSU 50-1-4
Record Dates: First submitted 2025-01-30; First posted 2025-02-05 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Analgesia; Vastus Lateralis Nerve Block; Lateral Femoral Cutaneous Nerve Block; Knee Surgeries
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vastus lateralis nerve block group (Experimental): Patients will receive vastus lateralis nerve block.
  Interventions: Drug: Vastus lateralis nerve block
- Lateral femoral cutaneous nerve block group (Experimental): Patients will receive lateral femoral cutaneous nerve.
  Interventions: Drug: Lateral femoral cutaneous nerve block

INTERVENTIONS:
Drug: Vastus lateralis nerve block — Patients received vastus lateralis nerve block with 5 ml of bupivacaine 0.5%.
  Other Names: Bupivacaine 0.5%
  Arms: Vastus lateralis nerve block group
Drug: Lateral femoral cutaneous nerve block — Patients received lateral femoral cutaneous nerve block with 5 ml of bupivacaine 0.5%.
  Other Names: Bupivacaine 0.5%
  Arms: Lateral femoral cutaneous nerve block group

SUMMARY:
This study aims to compare the analgesic efficacy and functional outcomes of blocking the nerve to the vastus lateralis (NVL) muscle versus the lateral femoral cutaneous nerve (LFCN).

DETAILED DESCRIPTION:
Knee surgeries are associated with significant postoperative pain, which can impede early mobilization and prolong recovery. Recent advancements in ultrasound-guided regional anesthesia have enabled more targeted nerve blocks, such as the blockade of the nerve to the vastus lateralis (NVL) and the lateral femoral cutaneous nerve (LFCN)

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status from I to III.
* Underwent knee surgeries under spinal anesthesia.

Exclusion Criteria:

* Pregnancy.
* Coagulopathy.
* Neuromuscular disorders.
* Hematological disorders.
* Mental disorders.
* History of multiple traumas or anesthesia drug allergies.
* Local skin infection at the block site.
* Body mass index (BMI) greater than 40.
* Opioid analgesics or abusing opioids.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-02-05 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-07-30 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment using the numeric rating scale (NRS) score (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS assessments will be conducted at the post-anesthesia care unit (PACU) and at 2, 4, 6, 12, 18, and 24 hours postoperatively.

SECONDARY OUTCOMES:
Time to first request for analgesia | 24 hours postoperatively
  The time to first request for analgesia will be recorded from the end of surgery till the first dose of morphine is administered.
Total morphine consumption | 24 hours postoperatively
  If the numeric rating scale (NRS) exceeded 3, rescue analgesia in the form of a 3 mg morphine bolus will be administered, to be repeated after 30 minutes if the pain persisted until the NRS dropped below 4.
Block performance time | Intraoperatively
  The block performance time will be recorded from the placement of the ultrasound probe to the removal of the needle after the injection of local anaesthetic.
Degree of patient satisfaction | 24 hours postoperatively
  The degree of patient satisfaction will be measured using a 5-point Likert scale (1 = extremely dissatisfied, 2 = unsatisfied, 3 = neutral, 4 = satisfied, 5 = extremely satisfied).
Length of hospital stay | Till the discharge from hospital (Up to one week).
  Length of hospital stay will be recorded from admission till discharge from the hospital.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as postoperative nausea and vomiting (PONV), respiratory depression, and local anesthetic (LA) toxicity will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Kafrelsheikh University, Kafr ash Shaykh, Kafrelsheikh, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.